# Statistical Analysis Plan

A prospective, multicenter, non-randomized, clinical outcomes study of the R30 Acetabular System in patients with degenerative hip disease

Number:

R3H01/02/01/2017

ST: 1103 Version: 3.0


# STATISTICAL ANALYIS PLAN (SAP)

#### **Study Details:**

| Protocol Version | 2.0 | Protocol Date | 01-Feb-2017 |
|------------------|-----|---------------|-------------|

#### **SAP Version Control:**

| SAP Status | Version 3.0, 06-Jun-2022 |
|------------------|--------------------------|
| Previous Version | version 1.0, 17-Nov-2020 |
| Number, Date | |

| Name and Title | Signature and Date / DocuSign Stamp |
|---|---|
| Babajide Olayinka<br>Senior Biostatistician<br>(Study Statistician) | DocuSigned by: Bahajidu Clayinka Signer Name: Babajide Olayinka Signing Reason: I am the author of this document Signing Time: 06-Jun-2022 20:58:52 BST 00FBF0F76B014495B7E2B2800B40F6AA |
| Sarah Megginson<br>Senior Biostatistician<br>Head of Global Biostatistics or<br>designee | DocuSigned by: Sanate Action Signer Name: Sarah Megginson Signing Reason: I have reviewed this document Signing Time: 06-Jun-2022 21:45:05 BST AB606B91C10B41909D3E0B2F7B357742 |

#### 

# **Statistical Analysis Plan**

A prospective, multicenter, non-randomized, clinical outcomes study of the R30 Acetabular System in patients with degenerative hip disease

Number:

R3H01/02/01/2017


### **Contents**

| STATISTICAL ANALYIS PLAN (SAP) | |
|-----------------------------------------------------|----|
| 1 List of Abbreviations | 4 |
| 2 Introduction | ε |
| 3 Study Design | ε |
| 4 Study Objectives | ε |
| 5 Study Endpoints | 7 |
| 5.1 Primary Endpoint | 7 |
| 5.2 Secondary Endpoint | 7 |
| 5.3 Safety Endpoints | 7 |
| 6 Statistical Considerations | 8 |
| 6.1 Determination of Sample Size | 8 |
| 6.2 Randomisation | 8 |
| 6.3 Interim Analysis | 8 |
| 7 Statistical Analysis | 8 |
| 7.1 General | |
| 7.2 Analysis Populations | g |
| 7.3 Handling of Missing, Incomplete and Repeat Data | g |
| 7.4 Derived Data | 10 |
| 7.5 Baseline Data | 14 |
| 7.6 Disposition Data | 14 |
| 7.7 Protocol Deviations | 14 |
| 7.8 Multiplicity | 15 |
| 7.9 Analysis of Primary Endpoint | 15 |
| 7.10 Analysis of Secondary Endpoints | 15 |
| 7.11 Analysis of Safety Endpoints | 16 |
| 7.12 Additional Analysis | 16 |
| 7.13 Other Data Summaries | 17 |

#### 

# **Statistical Analysis Plan**

A prospective, multicenter, non-randomized, clinical outcomes study of the R30 Acetabular System in patients with degenerative hip disease

Number:

R3H01/02/01/2017


| 7.14 Changes in Analysis Methods Specified in the Protocol | 1 | .7 |
|------------------------------------------------------------|---|----|
| 8 References | 1 | 8 |

#### 

# **Statistical Analysis Plan**

A prospective, multicenter, non-randomized, clinical outcomes study of the R30 Acetabular System in patients with degenerative hip disease

Number:

R3H01/02/01/2017

ST: 1103

Version: 3.0 

### 1 LIST OF ABBREVIATIONS

| ADE | Adverse Device Effect |
|-------|-------------------------------------------------|
| | Adverse Device Effect |
| ADL | Activity limitations daily living |
| AE | Adverse Event(s) |
| ASADE | Anticipated Serious Adverse Device Effect |
| CI | Confidence Interval |
| CRF | Case Report Form |
| DC | Discharge |
| DevD | Device Deficiency(ies) |
| FAS | Full Analysis Set |
| =U | Follow-Up |
| HHS | Harris Hip Score |
| HOOS | Hip Disability and Osteoarthritic Outcome Score |
| ISO | International Organization for Standardisation |
| LSLV | Last Subject Last Visit |
| MAR | Missing at Random |
| MMRM | Mixed Model Repeated Measure |
| N/A | Not Applicable |
| NICE | National Institute for Clinical Excellence |
| ODEP | Orthopaedic Data Evaluation Panel |
| OP | Operative |
| PP | Per-protocol Population |

#### 

# **Statistical Analysis Plan**

A prospective, multicenter, non-randomized, clinical outcomes study of the R30 Acetabular System in patients with degenerative hip disease

Number:

R3H01/02/01/2017


| Abbreviation | Definition |
|--------------|---------------------------------------------|
| QoL | Quality of Life |
| SADE | Serious Adverse Device Effect |
| SAE | Serious Adverse Event |
| SAF | Safety Analysis Set |
| SAP | Statistical Analysis Plan |
| TFL | Tables, Figures and Listing |
| UCLA | University of California, Los Angeles |
| USADE | Unanticipated Serious Adverse Device Effect |
| VAS | Visual Analogue Scale |

#### 

# **Statistical Analysis Plan**

A prospective, multicenter, non-randomized, clinical outcomes study of the R30 Acetabular System in patients with degenerative hip disease

Number:

R3H01/02/01/2017


### 2 INTRODUCTION

The following Statistical Analysis Plan (SAP) details the statistical considerations, including the data analysis methods, for the Study Protocol R3H01/02/01/2017 version 2.0/BNA. Related documents to this SAP are the Study Protocol, Case Report Form (CRF), and Table, Figure and Listing (TFL) Template Shells. This SAP is also an amendment to the previous finalized versions 1.0 and 2.0.

### 3 STUDY DESIGN

This is a multicenter prospective observational post-market clinical follow-up study that includes 512 patients who had a total hip replacement with the R3 Acetabular System and either cemented or cementless hip stem. The schedule of events is provided in Table 1.

Table 1. Study schedule of events

| Study Activity | Preop | Op | DC | 3M<br>(+/-<br>14d) | 1Y<br>(+/-<br>2m) | 3Y<br>(+/-<br>3m) | 5Y<br>(+/-<br>6m) | 7Y<br>(+/-<br>6m) | 10Y<br>(+/-<br>6m) |
|---|---|---|---|---|---|---|---|---|---|
| Inclusion/Exclusion | Χ | | | | | | | | |
| Informed Consent | Х | | | | | | | | |
| Demographics/Med<br>History | Х | | | | | | | | |
| Harris Hip Score | Χ | | | X | X | X | X | X | X |
| UCLA | Χ | | | Х | Х | X | X | X | Х |
| HOOS | Х | | | Х | Х | Х | Х | Х | Х |
| Radiograph Evaluation | | | X | | X* | X | X | X | X |
| Operative | | Χ | | | | | | | |
| Discharge | | | Х | | | | | | |
| Adverse Events | | Χ | Х | Х | Х | Х | Х | Х | Х |

<sup>\*</sup> Full pelvic overview

# **4 STUDY OBJECTIVES**

The objective of this study is to determine the long-term safety and effectiveness of the R3 Acetabular System by analysing the clinical, radiographic responses and the adverse event rates for

#### 

# **Statistical Analysis Plan**

A prospective, multicenter, non-randomized, clinical outcomes study of the R30 Acetabular System in patients with degenerative hip disease

Number:

R3H01/02/01/2017


patients undergoing primary total hip arthroplasty using the R3 Hip System (R3 Acetabular System). The study hypothesis is as follows: implant survivorship (Kaplan-Meier) (revision for any reason) of the R3 cup is at least 97% at 3 years, 95% at 5 years, 93% at 7 years, and 90% at 10 years follow-up.

### **5 STUDY ENDPOINTS**

# **5.1 Primary Endpoint**

The primary endpoint is implant survivorship at 10 years postoperatively.

### 5.2 Secondary Endpoint

Secondary endpoints include the following:

- Implant survivorship of the acetabular/cup at 10 years postoperatively
- Modified Harris Hip Score (mHHS)
- Hip disability and Osteoarthritis Outcome Score (HOOS)
- University of California, Los Angeles (UCLA) Rating
- Radiographic evaluation
- Patient Satisfaction

### **5.3 Safety Endpoints**

The safety endpoints are as follows:

- Incidence of Adverse Events by International Organization for Standardization (ISO) classifications
- Incidence of AEs by severity,
- o Incidence of AEs by relationship to study device,
- Incidence of serious adverse events (SAEs),
- o Incidence of Serious Adverse Device Effects (SADEs),
- o Incidence of Unanticipated Serious Adverse Device Effects (USADEs),
- Incidence of Anticipated Serious Adverse Device Effects (ASADEs),
- o Incidence of procedure-and or device related events,

#### 

# **Statistical Analysis Plan**

A prospective, multicenter, non-randomized, clinical outcomes study of the R30 Acetabular System in patients with degenerative hip disease

Number:

R3H01/02/01/2017

ST: 1103

Version: 3.0 

o Listing of revisions and components revised.

### **6 STATISTICAL CONSIDERATIONS**

### 6.1 Determination of Sample Size

The target enrollment during this study was 500 patients however 512 subjects have been enrolled. This number of patients leads to representative results with a greater precision of the survival rates, i.e. small confidence intervals.

The sample size is large enough to satisfy pseudo-regulatory requirements set-forth in individual European countries such as the Orthopaedic Data Evaluation Panel<sup>1</sup> (ODEP) and the National Institute for Clinical Excellence (NICE) requirements<sup>2</sup>. According to the ODEP criteria for categorizing products in relation to NICE's long-term benchmarks for hip replacements, a level A study (strongest evidence) requires an initial cohort of 500 patients or more.

### 6.2 Randomisation

Not applicable.

### 6.3 Interim Analysis

Not applicable as LSLV has been performed.

### **7 STATISTICAL ANALYSIS**

### 7.1 General

Smith+Nephew's Global Biostatistics group will conduct the statistical analysis for this study. Unless otherwise stated, all significance tests and hypothesis testing will be two-sided, performed at the 5% significance level. Resulting p-values will be quoted and 95% two-sided confidence intervals will be generated where appropriate. All p-values will be rounded to three decimal places, p-values less than 0.001 will be presented as '<0.001' in all tables.

#### 

# **Statistical Analysis Plan**

A prospective, multicenter, non-randomized, clinical outcomes study of the R30 Acetabular System in patients with degenerative hip disease

Number:

R3H01/02/01/2017


Where data summaries are specified, categorical and ordinal variables will be summarized with frequencies and percentages. Continuous variables will be summarized with the following summary statistics: number of observations, mean, median, standard deviation, minimum and maximum values. All analyses will be performed in SAS 9.4 (or later).

### 7.2 Analysis Populations

The following are the analysis populations used in summarizing all tables:

#### Safety Analysis Population (SAF)

This will include all subjects (Hips) enrolled and implanted with the study device in the study.

#### Full Analysis Set (FAS)

The FAS population will include all subjects (Hips) in the SAF with at least one postoperative assessment on any of the Patient Reported Outcome Measures (PROMs).

#### Per Protocol (PP) Population

The PP population will include all subjects (Hips) in FAS, who have no significant protocol deviations and satisfy all study eligibility criteria and the inclusion/exclusion criteria. Significant protocol deviations leading to removal from the PP population will be determined and finalized prior to the final analyses at 10 years. The final assignment of a subject to the PP population will be established after all protocol deviations have been reviewed and evaluated. Subjects excluded from the PP will be documented/listed together with their reason(s) for exclusion.

# 7.3 Handling of Missing, Incomplete and Repeat Data

For the primary endpoint, subjects with hips that are prematurely discontinued from the study due to death or loss to follow-up would be censored on the last known date on-study.

Specific instructions for handling missing PROMs is described in Section 7.4. If  $\geq$  10% of postoperative UCLA, HOOS or HHS scores at more than 2 of the postoperative follow-up time points are missing, only their observed data will be summarized using the change from preoperative to each postoperative time point as the endpoints of interest.

#### 

# **Statistical Analysis Plan**

A prospective, multicenter, non-randomized, clinical outcomes study of the R30 Acetabular System in patients with degenerative hip disease

Number:

R3H01/02/01/2017


#### 7.4 Derived Data

#### Body Mass Index (BMI)

- o BMI =  $\{(Weight in kg)/(Height in m)^2\}$ , if units are in kg for weight and m for height OR;
- o BMI = {(Weight in lbs)x703.07))/(Height in inches) $^2$ }, if units are in lbs for weight and inches for height (Adjustments made to formula to standardize BMI unit to kg/m $^2$ ).

#### Change from baseline

Change from baseline (preoperative) scores to postoperative time points (i.e. Visit<sub>i</sub>) for all pertinent endpoints would be calculated at follow-up visits as follows: Postoperative visit<sub>i</sub> score – preoperative score.

#### Hip Disability and Osteoarthritis Outcome Score (HOOS)

The HOOS consists of 3 subscales; Pain, Stiffness and Function in daily living (ADL). Five standardized answer options are given and each question gets a score from 0 to 4. The detailed information is showed in Table 2. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) for each subscale will be calculated as:

HOOS pain = 100 - AVERAGE (P1:P5)\* 100/4HOOS Stiffness = 100 - AVERAGE (S4:S5)\* 100/4HOOS ADL = 100 - AVERAGE (A1:A17)\* 100/4

#### Table 2 HOOS Domain Questionnaire and Scores

| HOOS Item # | HOOS Items (Individual item scores 0-4, with None = 0; Mild = 1; Moderate = |
|---|---|
| | 2; Severe = 3; Extreme = 4) |
| Pain (score range 0-20) | |
| P1 | Walking on a flat surface? |
| P2 | Going up or down stairs? |
| Р3 | At night while in bed? |
| P4 | Sitting or lying? |
| P5 | Standing upright? |
| Stiffness (score range 0-8) | |
| S4 | Severity of stiffness after first wakening in the morning? |
| S5 | Severity of stiffness after sitting/lying/resting later in the day? |
| ADL (score range 0-68) | |
| A1 | Descending stairs? |
| A2 | Ascending stairs? |

#### 

# **Statistical Analysis Plan**

A prospective, multicenter, non-randomized, clinical outcomes study of the R30 Acetabular System in patients with degenerative hip disease

Number:

R3H01/02/01/2017

ST: 1103

Version: 3.0 

| A3 | Rising from sitting? |
|-----|-------------------------------------|
| A4 | Standing? |
| A5 | Bending to floor/pick up an object? |
| A6 | Walking on flat surface? |
| A7 | Getting in/out of car? |
| A8 | Going shopping? |
| A9 | Putting on socks/stockings? |
| A10 | Rising from bed? |
| A11 | Taking off socks/stockings? |
| A12 | Lying in bed? |
| A13 | Getting in/out of bath/shower? |
| A14 | Sitting? |
| A15 | Getting on/off toilet? |
| A16 | With heavy domestic duties? |
| A17 | With light domestic duties? |

If there are some missed answers, then the following rule will be followed.

- 1. For each subscale, if there are at least 50% of the items are answered, then we will calculate the subscale mean score as showed in Table 3.
- 2. For each subscale, if more than 50% of items are missed, then we will not calculate subscale mean score.
- 3. Subscale scores will be calculated independently, i.e. if a particular subscale is not valid, the results from the other subscale will still be calculated if available.

Table 3 Number of items needed for each subscale

| SubDomain | # of items need to for calculation subscale mean score |
|-----------|--------------------------------------------------------|
| Pain | 3 |
| Stiffness | 1 |
| ADL | 9 |

#### Modified Harris Hip Score (HHS)

The mHHS includes a modification to the Harris Hip Score: the "Distance Walked" section of the Harris Hip Score was modified to replace the number of blocks with actual distances since the term "blocks" is not commonly used as a measurement of distance in Europe.

Table 4 displays the algorithms used for scoring each of the 10 items (components) of the mHHS as well as the domains (pain, function, AoD and ROM) of the mHHS and total mHHS.

Table 4. modified Harris Hip Score (HHS) scores per item and domain

#### 

# **Statistical Analysis Plan**

A prospective, multicenter, non-randomized, clinical outcomes study of the R30 Acetabular System in patients with degenerative hip disease

Number:

R3H01/02/01/2017


| | | Likely scores | Domains (Range of |
|---|---|---|---|
| Item | Original Response | per Item | Scores) |
| Pain | None or ignores it | 44 | Pain Domain (0 to |
| | Slight, minimal, no compromise in activities | 40 | |
| | Mild pain, no effect on average activities, rarely moderate pain with unusual activity; may take aspirin | 30 | |
| | Moderate pain; tolerable but makes concessions to pain. Some limitation of ordinary activity or work. May require occasional pain medication stronger than aspirin | 20 | |
| | Marked pain, serious limitation of activities | 10 | |
| | Totally disabled, crippled, pain in bed, bedridden | 0 | |
| Limp | None | 11 | Function Domain ( |
| | Slight | 8 | to 47) |
| | Moderate | 5 | |
| | Severe | 0 | {Sum of all items within subdomain |
| Support | None | 11 | |
| | Single cane for long walks | 7 | |
| | Single cane most of the time | 5 | |
| | One crutch | 3 | |
| | Two canes | 2 | |
| | Two crutches or not able to walk | 0 | |
| Distance walked | Unlimited | 11 | |
| | Six blocks | 8 | |
| | Daily shopping | 5 | |
| | Indoors only | 2 | |
| | Bed and chair only | 0 | |
| Sitting | Comfortably in ordinary chair | 5 | |
| | On a high chair for 30 minutes | 3 | |
| | Unable to sit comfortably in any chair | 0 | |

#### 

# **Statistical Analysis Plan**

A prospective, multicenter, non-randomized, clinical outcomes study of the R30 Acetabular System in patients with degenerative hip disease

Number:

R3H01/02/01/2017


| Stairs | Public | Yes, possible | 1 | ] |
|---|---|---|---|---|
| No, unable 0 | | res, possible | ı | |
| Normally without using a railing | transportation | No unable | 0 | |
| Normally using a railing | | No, unable | U | |
| In any manner | Stairs | Normally without using a railing | 4 | - |
| Unable to do stairs 0 | | Normally using a railing | 2 | |
| Socks/Shoes With ease With difficulty 2 Unable 0 | | In any manner | 1 | |
| With difficulty | | Unable to do stairs | 0 | |
| Unable | Socks/Shoes | With ease | 4 | - |
| Unable | | With difficulty | 2 | |
| Movement = ABD+ADD-ABD_ZERO N/A Rotation = ER+IR-ER_ZERO N/A | | • | | |
| Movement = ABD+ADD-ABD_ZERO N/A Rotation = ER+IR-ER_ZERO N/A | Range of Motion | Flexion = FLEX+EXT-FLEX_ZERO | N/A | |
| ROM subscore Flexion+Movement+Rotation 0 to 29 | | Movement = ARD+ADD-ARD 7EPO | NI/A | |
| ROM subscore Flexion+Movement+Rotation | | | | |
| Domain (0 to 5)) 0 to 29 30 to 59 60 to 99 2 100 to 159 360 to 209 ≥ 209 5 Leg Length Difference (in mm) Ipsilateral longer (LL_DIF_LONG) Ipsilateral shorter (LL_DIF_SHORT) N/A Absence of Deformity (AOD) 31) AND (ABD_ZERO = . OR ABD_ZERO < 11) AND (ER_ZERO = . OR ER_ZERO < 11) AND LL_DIF_LONG < 33 AND LL_DIF_SHORT < 33 THEN AODScore = 4 Total HHS Sum of all Sum of all Sum of all | | Rotation - ERTIR-ER_ZERO | N/A | |
| 30 to 59 60 to 99 2 100 to 159 3 160 to 209 4 ≥ 209 5 Leg Length Difference (in mm) Ipsilateral longer (LL_DIF_LONG) Ipsilateral shorter (LL_DIF_SHORT) N/A Absence of Deformity (AOD) IF (FLEX_ZERO = . OR FLEX_ZERO < 0 or 4 Deformity (AOD) 31) AND (ABD_ZERO = . OR ABD_ZERO < 11) AND (ER_ZERO = . OR ER_ZERO < 11) AND LL_DIF_LONG < 33 AND LL_DIF_LONG < 33 THEN AODScore = 4 Total HHS Sum of all Sum of all Sum of all | ROM subscore | Flexion+Movement+Rotation | | _ |
| 60 to 99 | | 0 to 29 | 0 | |
| 100 to 159 160 to 209 ≥ 209 Leg Length Difference (in mm) Ipsilateral longer (LL_DIF_LONG) N/A Ipsilateral shorter (LL_DIF_SHORT) N/A N/A Ipsilateral shorter (LL_DIF_SHORT) N/A N/A Ipsilateral shorter (LL_DIF_SHORT) N/A N/A | | 30 to 59 | 1 | |
| 160 to 209 ≥ 209 5 Leg Length Difference (in mm) Ipsilateral longer (LL_DIF_LONG) Ipsilateral shorter (LL_DIF_SHORT) N/A Absence of Deformity (AOD) IF (FLEX_ZERO = . OR FLEX_ZERO < 0 or 4 Absence of ABD_ZERO < 11) AND (ER_ZERO = . OR ER_ZERO < 11) AND LL_DIF_LONG < 33 AND LL_DIF_SHORT < 33 THEN AODScore = 4 Total HHS Sum of all Sum of all Sum of all | | 60 to 99 | 2 | |
| ≥ 209 5 Leg Length None N/A Difference (in mm) Ipsilateral longer (LL_DIF_LONG) N/A Ipsilateral shorter (LL_DIF_SHORT) N/A Absence of Deformity (AOD) IF (FLEX_ZERO = . OR FLEX_ZERO < 0 or 4 OR ER_ZERO < 11) AND (ER_ZERO = . OR ABD_ZERO = . OR ER_ZERO < 11) AND (ER_ZERO = . OR ER_ZERO < 11) AND LL_DIF_LONG < 33 AND LL_DIF_SHORT < 33 THEN AODScore = 4 | | 100 to 159 | 3 | |
| Leg Length None N/A Difference (in mm) Ipsilateral longer (LL_DIF_LONG) N/A Ipsilateral shorter (LL_DIF_SHORT) N/A Absence of IF (FLEX_ZERO = . OR FLEX_ZERO < 0 or 4 Deformity (AOD) 31) AND (ABD_ZERO = . OR ABD_ZERO < 11) AND (ER_ZERO = . OR ER_ZERO < 11) AND LL_DIF_LONG < 33 AND LL_DIF_SHORT < 33 THEN AODScore = 4 Total HHS Sum of all Sum of all Sum of all | | 160 to 209 | 4 | |
| Ipsilateral longer (LL_DIF_LONG) N/A Ipsilateral shorter (LL_DIF_SHORT) N/A Absence of | | ≥ 209 | 5 | |
| Ipsilateral longer (LL_DIF_LONG) N/A Ipsilateral shorter (LL_DIF_SHORT) N/A Absence of | Lea Lenath | None | N/A | |
| Ipsilateral longer (LL_DIF_LONG) N/A | | | | |
| Ipsilateral shorter (LL_DIF_SHORT) N/A N/A | , | Ipsilateral longer (LL_DIF_LONG) | N/A | |
| Absence of | | · | | |
| Deformity (AOD) 31) AND (ABD_ZERO = . OR | | .poa.c.a. eec. ( <u></u> _eee., | ,, . | |
| ABD_ZERO < 11) AND (ER_ZERO = . OR ER_ZERO < 11) AND LL_DIF_LONG < 33 AND LL_DIF_SHORT < 33 THEN AODScore = 4 Total HHS Sum of all Sum of all domain | Absence of | IF (FLEX ZERO = . OR FLEX ZERO < | 0 or 4 | Absence of |
| ABD_ZERO < 11) AND (ER_ZERO = . OR ER_ZERO < 11) AND LL_DIF_LONG < 33 AND LL_DIF_SHORT < 33 THEN AODScore = 4 Total HHS Sum of all Sum of all domain | Deformity (AOD) | ` = | | <b>Deformity Domain</b> |
| OR ER_ZERO < 11) AND LL_DIF_LONG < 33 AND LL_DIF_SHORT < 33 THEN AODScore = 4 Total HHS Sum of all Sum of all domain | , | | | |
| LL_DIF_LONG < 33 AND LL_DIF_SHORT < 33 THEN AODScore = 4 Total HHS Sum of all Sum of all domain | | _ | | |
| LL_DIF_SHORT < 33 THEN AODScore = 4 Total HHS Sum of all Sum of all domain | | _ <i>,</i> | | |
| = 4 Total HHS Sum of all Sum of all domain | | | | |
| | Total UUC | | Cura of all | Cum of all domes!:- |
| TOPINE TAR SENTE DE PARTE MARIE MARI | I Olai MMS | | | |
| per subject | | | | scores per subject |
| per subject | | | per subject | |

#### 

# **Statistical Analysis Plan**

A prospective, multicenter, non-randomized, clinical outcomes study of the R30 Acetabular System in patients with degenerative hip disease

Number:

R3H01/02/01/2017

ST: 1103

Version: 3.0 

Note: The maximum possible score for the HHS is 100.

### 7.5 Baseline Data

The following preoperative, operative and demographic variables would be summarized using descriptive characteristics for continuous<sup>1</sup> or categorical<sup>2</sup> data as appropriate:

- Age<sup>1</sup> (in years),
- Sex² (males or females),
- Height<sup>1</sup> (in cm),
- Weight¹ (in kg),
- o BMI<sup>1</sup>
- Primary diagnosis<sup>2</sup>,
- Charnley classification<sup>2</sup>
- Surgical history ipsilateral<sup>2</sup>
- ASA Physical Status<sup>2</sup>
- Head, Size, Neck Length, Inlay Material, Inlay<sup>2</sup>
- Surgical Approach<sup>2</sup>

Variables summarized will not only be restricted to the above listed but all variables deemed pertinent and obtainable preoperatively and operatively.

# 7.6 Disposition Data

Hip accountability will be summarized by study visit (see Table 1 for visit schedule) for the number of hips that are theoretically due, subjects who died, hips that were revised, hips terminated from the study for any reason. Additional information will include but not limited to number of subjects presenting at each visit, number of hips expected at each visit and follow up rate.

### 7.7 Protocol Deviations

A listing of all protocol deviations encountered on-study will be summarized.

#### 

# **Statistical Analysis Plan**

A prospective, multicenter, non-randomized, clinical outcomes study of the R30 Acetabular System in patients with degenerative hip disease

Number:

R3H01/02/01/2017


# 7.8 Multiplicity

No adjustments for multiplicity are planned for this study.

### 7.9 Analysis of Primary Endpoint

The Kaplan-Meier survival estimate would be used to estimate implant survivorship. Time to device revision will be the endpoint of interest to estimate the implant survivorship. Implant survival time (in months) is computed as: (Event Date – Operative Date+1)/30.4375.

Implanted hips that continue until study completion without an on-study revision will be censored at their last known date of participation in the study. Any premature hip discontinuation from study due to a subject's death or any other reason will be censored on the date of this discontinuation. A subject who is lost to follow-up will be censored at the subject's last known contact date. The Cumulative proportion of implant survivorship at 36 months (3-year), 60 months (5 years), 84 months (7 years) and 120 months (10 years) will be estimated and displayed accordingly. These Kaplan-Meier estimates will be provided with their corresponding two-sided 95% Confidence Intervals (CIs). If feasible, Kaplan-Meier survival graphs will be displayed to graphically illustrate implant survivorship over the study duration.

For the a-priori protocol-specified hypothesis, if the lower bound of 95% two-sided CIs at 3 years, 5 years, 7 years and 10 years are not less than 97%, 95%, 93% and 90% respectively, then we conclude that implant survivorship of the R3 cup is at least 97% at 3 years. 95% at 5 years, 93% at 7 years, and 90% at 10 years follow-up respectively.

The primary endpoint analysis will be performed on the FAS population. As sensitivity analysis, the same analysis will be performed on the PP population.

# 7.10 Analysis of Secondary Endpoints

HOOS sub-scores, HHS (and the its subscores) and UCLA would be summarized using
descriptive summary characteristics for continuous variables at the preoperative and all
postoperative time points. Changes from the preoperative (baseline) to subsequent
postoperative visit(s) would also be summarized using descriptive statistics for continuous

#### 

# **Statistical Analysis Plan**

A prospective, multicenter, non-randomized, clinical outcomes study of the R30 Acetabular System in patients with degenerative hip disease

Number:

R3H01/02/01/2017


variables. Mixed Model Repeated Measures (MMRM) with a missing at random (MAR) assumption to account for the pattern of missing longitudinal data would be used to analyze the Patient Reported Outcome Measures (PROMs) to compare the scores between the preoperative and postoperative visit time points. The model will include fixed effect term for visit. The Kenward Rogers denominator degrees of freedom would be used coupled with a specification for an unstructured covariance matrix. The test of any of the comparisons between the preoperative and postoperative visits will be concluded to be statistically significant if p < 0.05. Model-based Means or Least Square (LS) Means for all visits as well as the differences between each postoperative versus the preoperative visit and their 95% two-sided Confidence Intervals (CI) would be presented. Should greater than 10% of any of the PROMs data on at least at two of the postoperative timepoints be missing, MMRM would not be used.

• For radiographic findings, patient satisfaction and Trendelenburg, descriptive summary statistics for categorical variables such as frequency (n) and percentage (%) will be presented by visit.

The secondary endpoint analysis will be performed only on the FAS population.

### 7.11 Analysis of Safety Endpoints

An overall summary AE table that would summarize as number (n) and percentages (%), the overall incidence according to subjects (and hips) with at least one AE; subjects (and hips) with at least one AE by worst severity (mild, moderate, or severe), by worst outcome (resolved, ongoing/unresolved, death or removal/revision of components), worse relatedness to device, SAEs, ADEs, SADEs and, USADEs. Classification of AEs would also be summarized using ISO classifications. A data listing with all AEs (and their classifications) reported on-study will be presented. Finally, the incidence of device-and/or procedure related AE by their type will be presented too.

### 7.12 Additional Analysis

Type of R3 bearing would be classified into meaningful subgroups by the Clinical Strategy team using Head/Inlay/Inlay Material available in the database. Implant survivorship would subsequently be summarized exploratorily for each of the classified subgroup of the R3 bearing (head/inlay: i.e. Biolox delta ceramic-on-ceramic, Biolox forte ceramic-on-ceramic, Oxidized zirconium-on-

#### 

# **Statistical Analysis Plan**

A prospective, multicenter, non-randomized, clinical outcomes study of the R30 Acetabular System in patients with degenerative hip disease

Number:

R3H01/02/01/2017


crosslinked polyethylene, Ceramic-on-crosslinked polyethylene, Metal-on-crosslinked polyethylene and Metal-on-metal) using Kaplan-Meier survival methods as described in Section 7.9.

The analysis population for these analyses would be the FAS population.

#### 7.13 Other Data Summaries

Not applicable.

### 7.14 Changes in Analysis Methods Specified in the Protocol

The protocol-specified hypothesis is now more carefully elucidated in this SAP.

The primary analysis population of the primary endpoint is now specified to the based on the FAS population.

After consultation between key study stakeholders, it was determined that the additional COVID-related analyses previously included in SAP final version 1.0 would be of negligible-to-no impact on the results and therefore this is removed from this amendment.

Additional exploratory analysis of the primary endpoint by head/inlay material was added on request by Clinical Strategy.

#### 

# **Statistical Analysis Plan**

A prospective, multicenter, non-randomized, clinical outcomes study of the R30 Acetabular System in patients with degenerative hip disease

Number:

R3H01/02/01/2017


#### 8 REFERENCES

- 1. ODEP criteria for categorizing data in relation to NICE's benchmarks. *Orthopaedic Data Evaluation Panel*. 2005.
- 2. NICE. Guidance on the selection of prostheses for primary total hip replacement. *Technology Appraisal Guidance No. 2. National Institute for Health and Clinical Excellence*. 2000.

#### 

#### **Certificate Of Completion**

Envelope Id: 0184139470EB41089627E0E2EAE09C0F

Subject: Please DocuSign: 2022 06.06 R3 EU Pro R11019\_SAP Observational Study Final V3.0.docx

Source Envelope:

Document Pages: 18 Signatures: 2 Certificate Pages: 2 Initials: 0 Babajide Olayinka

AutoNav: Enabled

Envelopeld Stamping: Enabled

Time Zone: (UTC) Dublin, Edinburgh, Lisbon, London

**Envelope Originator:** 

TJ Smith & Nephew Limited

101 Hessle Road Hull, Hull HU3 2BN

Status: Completed

Babajide.olayinka@smith-nephew.com

IP Address: 204.9.32.4

Sent: 06-Jun-2022 | 20:49

Viewed: 06-Jun-2022 | 20:57

Signed: 06-Jun-2022 | 20:58

Sent: 06-Jun-2022 | 20:49

Viewed: 06-Jun-2022 | 21:44

Signed: 06-Jun-2022 | 21:45

#### **Record Tracking**

Status: Original

06-Jun-2022 | 20:47

Holder: Babajide Olayinka

Babajide.olayinka@smith-nephew.com

# **Timestamp**

Location: DocuSign

**Signer Events** Babajide Olayinka

babajide.olayinka@smith-nephew.com

Biostatistics/Data Manager 2

Smith & Nephew

Security Level: Email, Account Authentication

(Required)

Babajide Olayinka

Signature Adoption: Pre-selected Style

Signed by link sent to

babajide.olayinka@smith-nephew.com

Signature ID:

Signature

00FBF0F7-6B01-4495-B7E2-B2800B40F6AA

Using IP Address: 204.9.32.4

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab): I am the author of this document

#### **Electronic Record and Signature Disclosure:**

Not Offered via DocuSign

Sarah Megginson

Sarah.Megginson@smith-nephew.com

Biostatistics/Data Analyst 3

Smith & Nephew

Security Level: Email, Account Authentication

(Required)

Sarah Megginson

Signature Adoption: Pre-selected Style

Signed by link sent to

Sarah.Megginson@smith-nephew.com

Signature ID:

AB606B91-C10B-4190-9D3E-0B2F7B357742

Using IP Address: 216.222.214.6

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab): I have reviewed this document

#### **Electronic Record and Signature Disclosure:**

Not Offered via DocuSign

In Person Signer Events

Signature **Timestamp** 

**Editor Delivery Events** Status **Timestamp** 

**Agent Delivery Events Status Timestamp** 

| Intermediary Delivery Events | Status | Timestamp |
|---|---|---|
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 06-Jun-2022 20:49 |
| Certified Delivered | Security Checked | 06-Jun-2022 21:44 |
| Signing Complete | | 00 1 2000 1 24.45 |
| oighing complete | Security Checked | 06-Jun-2022 21:45 |
| Completed | Security Checked Security Checked | 06-Jun-2022 21:45<br>06-Jun-2022 21:45 |